CLINICAL TRIAL: NCT02788916
Title: A Retrospective Study of Clinical, Phenotypic and Genetic Factors of Peripheral T-Cell Lymphomas in the Spanish Population
Brief Title: A Retrospective Study of Clinical, Phenotypic and Genetic Factors of Peripheral T-Cell Lymphomas
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brentuximab-5012; TAK-HEM-2015-01 (Registry Identifier: AEMPS)
Record Dates: First submitted 2016-05-23; First posted 2016-06-02 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Initial tumor biopsies and histological preparations, filed and previously anonymized, will be assessed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Assessment of tumor biopsies and histological preparations of participants diagnosed with peripheral T-cell lymphoma (PTCL) in the six years between 01 January 2008 and 31 December 2013 will be performed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study is to establish the distribution of peripheral T-cell lymphocyte (PTCL) subtypes by re-analysis and re-classification of samples according to the 2008 World Health Organization (WHO) classification of lymphoid neoplasms.

DETAILED DESCRIPTION:
This study is a retrospective, non-interventional and, post-authorization observational study of other designs (PAS-OD).

This multicenter trial will be conducted in Spain. Retrospective review of medical records and initial tumor biopsies of participants diagnosed with PTCL in the period of 6 years between 01/01/2008 and 31/12/2013 will be performed. Initial tumor biopsies and histological preparations, filed and previously anonymized, will be sent to the central laboratory for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with PTCL in the six years between 01/01/2008 and 31/12/2013.
* Availability of initial tumor biopsy diagnosis in paraffin block (node or core biopsy of 16-18mm).
* PTCL subtypes permitted by WHO 2008 classification of lymphoid neoplasms:

  * Natural killer/ T-lymphocytes (NK /T-cell) lymphoma extranodal nasal type
  * Enteropathic T-cell lymphoma
  * Hepatosplenic T-cell lymphoma
  * Peripheral T-cell lymphoma, not otherwise specified
  * Angioimmunoblastic T-cell lymphoma
  * Anaplastic large cell lymphoma, Anaplastic lymphoma kinase positive (ALK)+
  * Anaplastic large cell lymphoma, ALK-

Exclusion Criteria:

• Participants with an unavailable history (lost, empty or not recoverable).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with PTCL in the six years between 01 January 2008 and 31 December 2013 in the participating sites.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Distribution of Peripheral T-cell Lymphoma (PTCL) Subtypes | Up to 6 months
  Distribution of PTCL subtypes by re-analysis and re-classification of samples according to the 2008 WHO classification of lymphoid neoplasms will be estimated.

SECONDARY OUTCOMES:
Percentage of Participants with Each Subtypes of PTCL | Up to 6 months
  Percentage of participants with each subtypes of PTCL according to the WHO 2008 classification of lymphoid neoplasms will be reported.
Rate of Discrepancy Between the Initial Diagnosis and Re-analysis and Re-classification | Up to 6 months
  Rate of discrepancy between the initial diagnosis of PTCL in participants and diagnosis by re-analysis and re-classification according to the WHO 2008 classification will be determined.
Expression of Cluster of Differentiation 30 (CD30) by Immunohistochemistry and Quantitative Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) in Different Subtypes of PTCL | Up to 6 months
  Expression of CD30 by immunohistochemistry and quantitative RT-PCR in different subtypes of PTCL will be determined.
Correlation Between the Expression of CD30 and Lymphoid Lineage | Up to 6 months
  Markers of T and B cells will be used in order to determine if CD30 expression occurs in tumor cells or other B-lineage.
Correlation Between the Expression of CD30, Prognostic Indices Used In PTCL and Survival | Up to 6 months
  Survival includes progression free survival: period from date of start of treatment until tumor progression or death, whichever occurs first. Overall survival: period from date of diagnosis to the date of death.
Classification of Peripheral T-cell Lymphoma | Up to 6 months
  The PTCL is classified according to the expression of CD30 and T-Cell Receptor ß (TCRß) and T-Cell Receptor γ (TCRγ) by immunohistochemistry (IHC).
T-cell Clonality in PTCL | Up to 6 months
  Analysis of T-cell clonality in PTCL will be performed. Clonality defines the profile of gene rearrangement of T cell receptor and allow establishing whether proliferation is monoclonal.
Correlation Between Most frequent Mutations and Clinical, Phenotypic Factors | Up to 6 months
  Distribution of the most frequent mutations in tumors and its correlation with clinical and phenotypic factors will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- Spain (10):
  - Santiago de Compostela, A Coruna
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Córdoba, Cordoba
  - Madrid, Madrid
  - Majadahonda, Madrid
  - Oviedo, Oviedo
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Valencia, Valencia